CLINICAL TRIAL: NCT01337973
Title: Impact of Interventions to Reduce Violence and Substance Abuse Among VA Patients
Brief Title: Preventing Violence Among Veterans in Substance Use Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 09-333; HX000294 (Other Grant/Funding Number: VA Merit Review Grant)
Record Dates: First submitted 2010-12-17; First posted 2011-04-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Aggression; Substance-Related Disorders
Keywords: violence; aggression; Substance-Related Disorders; Alcohol-Related Disorders; Drug-Related Disorders
MeSH Terms: conditions — Aggression; Substance-Related Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: MI-CBT (Experimental): MI-CBT (six sessions during acute treatment phase integrating motivational interviewing and cognitive behavioral approaches)
  Interventions: Behavioral: MI-CBT
- Arm 2: MI-CBT+CC (Experimental): MI-CBT+CC (acute phase MI-CBT intervention plus a subsequent 12-week phone based continuing care counseling intervention)
  Interventions: Behavioral: MI-CBT+CC
- Arm 3: E-TAU (Active Comparator): E-TAU (enhanced treatment as usual - includes brief session and provision of resources)
  Interventions: Behavioral: E-TAU

INTERVENTIONS:
Behavioral: MI-CBT — Six individual psychotherapy sessions during the acute substance use disorder treatment phase integrating motivational interviewing and cognitive behavioral approaches
  Arms: Arm 1: MI-CBT
Behavioral: MI-CBT+CC — Acute phase MI-CBT intervention plus a subsequent 12-week phone based continuing care counseling intervention
  Arms: Arm 2: MI-CBT+CC
Behavioral: E-TAU — Enhanced Treatment as Usual
  Arms: Arm 3: E-TAU

SUMMARY:
The purpose of this study is to examine the impact on both clinical (violence and substance use) outcomes and health services use (substance use disorder and mental health treatment) compared to standard SUD treatment (enhanced treatment as usual) of

1. an integrated Motivational Interviewing-Cognitive Behavioral Therapy (MI-CBT) violence prevention treatment intervention delivered during the 8-week early substance use disorder treatment phase; and
2. MI-CBT plus a continuing care (CC) intervention for the 3-month continuing care period following the early treatment phase MI-CBT+CC).

The study will provide important new information regarding the role and relative impact of both early treatment and continuing care interventions designed to impact substance use and violence, and whether combining such interventions yields additional benefits.

DETAILED DESCRIPTION:
Objective: Rates of violence in Substance Use Disorder (SUD) treatment samples often exceed 50%, with studies showing rates of past-year violence >70% when considering violence occurring with either intimate partners or others. Violence has numerous costs to Veterans and their families, in terms of physical (e.g., injuries) and psychosocial problems (mental health, legal problems, marital problems, poorer functioning for their children, etc.). To date, only one treatment approach (Behavioral Couples Therapy - BCT) has been established that reduces both substance use and violence, and BCT focuses exclusively on the couples' relationship. Given that a small proportion of Veterans in SUD treatment have a partner willing or able to attend treatment, and that a substantial amount of violence occurs with non-partners, there is a clear need for interventions that do not require partner participation and focus on violence and relapse prevention more generally. Based on prior findings, new intervention approaches targeting the use of violence prevention skills and means of sustaining substance use remission are needed.

The primary objectives of this study are to examine the impact on both substance use and violence outcomes of:

1. an acute treatment phase integrated Motivational Interviewing-Cognitive Behavioral Treatment intervention (MI-CBT); and
2. MI-CBT plus a violence and substance use prevention Continuing Care intervention (MI-CBT+CC) intervention.

Research Plan: Participants will be randomized to one of three conditions: MI-CBT, MI-CBT+CC or an enhanced treatment as usual (E-TAU) control condition with follow-up interviews targeting violence and substance use outcomes at 3, 6 and 12-months. The MI-CBT intervention involves six individual sessions delivered during the acute SUD treatment phase, combines Motivational Interviewing (MI) and CBT approaches targeting violence and substance use, and has been developed, piloted and refined by the investigators. The MI-CBT+CC intervention includes acute phase MI-CBT plus weekly telephone sessions for an additional 3-month period, and is designed to address both post-treatment violence and substance use through facilitating SUD remission and use of violence prevention skills. The MI-CBT+CC intervention is adapted from a continuing care intervention shown to help consolidate and maintain gains made in treatment.

Methods: Veterans with substance use disorders will be recruited from the Substance Abuse Clinic (SAC) at the VA Ann Arbor Healthcare system. Approximately 855 Veterans enrolling in SAC will be consented and screened, and those screening positive for severe and recent violence (~30%) and meeting other project inclusion/exclusion criteria will be eligible for participation in the randomized controlled trial (n = 210). The clinical interventions will be delivered by master's level clinicians, who will be monitored and supervised by licensed psychologists. Primary dependent measures (violence, substance use) will be measured at baseline and follow-up interviews, and the impact of the interventions on services use during the follow-up period also will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Participants with severe and recent violence (i.e., injuring another person in the past year) will be eligible for the RCT.
* Eligible patients also will meet DSM-IV criteria for either alcohol or illicit drug (e.g., cocaine, marijuana, opiates, etc.) abuse/dependence.
* The study will include those with comorbid mood and/or anxiety problems (e.g., depression, PTSD and other anxiety disorders), whether or not on medication at the point of recruitment, with the exception of those who have schizophrenia and/or are mentally incompetent (e.g., unable to provide informed consent).
* A brief mental status screen will with an established cutoff will be required for competency.

Exclusion Criteria:

* Participants who are suicidal (ideation, intent and plan) at the point of recruitment will not be enrolled in the study. Rather, research staff will inform clinical staff at the study site if a potential participant is currently suicidal.
* Participants who report transient suicidal ideation but no intent or plan will be eligible to participate.
* As noted, individuals with schizophrenia and/or who are mentally incompetent to consent for participation will be excluded. Finally, participants who live outside the study catchment area (i.e., a 45 mile radius of the VA Ann Arbor Healthcare System) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T. Chermack, PhD MA BA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis AK, Bonar EE, Ilgen MA, Walton MA, Perron BE, Chermack ST. Factors associated with having a medical marijuana card among Veterans with recent substance use in VA outpatient treatment. Addict Behav. 2016 Dec;63:132-6. doi: 10.1016/j.addbeh.2016.07.006. Epub 2016 Jul 8. PMID 27475408
- [Background] Bennett DC, Morris DH, Sexton MB, Bonar EE, Chermack ST. Associations between posttraumatic stress and legal charges among substance using veterans. Law Hum Behav. 2018 Apr;42(2):135-144. doi: 10.1037/lhb0000268. Epub 2017 Oct 26. PMID 29072473
- [Background] Anderson RE, Bonar EE, Walton MA, Goldstick JE, Rauch SAM, Epstein-Ngo QM, Chermack ST. A Latent Profile Analysis of Aggression and Victimization Across Relationship Types Among Veterans Who Use Substances. J Stud Alcohol Drugs. 2017 Jul;78(4):597-607. doi: 10.15288/jsad.2017.78.597. PMID 28728642
- [Background] Davis AK, Bonar EE, Goldstick JE, Walton MA, Winters J, Chermack ST. Binge-drinking and non-partner aggression are associated with gambling among Veterans with recent substance use in VA outpatient treatment. Addict Behav. 2017 Nov;74:27-32. doi: 10.1016/j.addbeh.2017.05.022. Epub 2017 May 20. PMID 28570911
- [Background] Buchholz KR, Bohnert KM, Sripada RK, Rauch SA, Epstein-Ngo QM, Chermack ST. Associations between PTSD and intimate partner and non-partner aggression among substance using veterans in specialty mental health. Addict Behav. 2017 Jan;64:194-199. doi: 10.1016/j.addbeh.2016.08.039. Epub 2016 Aug 31. PMID 27636157
- [Result] Chermack ST, Bonar EE, Goldstick JE, Winters J, Blow FC, Friday S, Ilgen MA, Rauch SAM, Perron BE, Ngo QM, Walton MA. A randomized controlled trial for aggression and substance use involvement among Veterans: Impact of combining Motivational Interviewing, Cognitive Behavioral Treatment and telephone-based Continuing Care. J Subst Abuse Treat. 2019 Mar;98:78-88. doi: 10.1016/j.jsat.2019.01.001. Epub 2019 Jan 4. PMID 30665608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from June 2012-June 2015 from outpatient VA mental health programs (Substance Use Disorder, Substance use Disorder Intensive Outpatient, General Mental Health).
Pre-assignment Details: Of 1097 eligible for screening, 183 refused participation (17%), 75 (7%) were missed and 839 completed the screening assessment. Of those completing screening, 639 were not eligible for the RCT and 20 refused further participation. Thus, 180 out of 200 eligible veterans (90%) were randomized to one of the three treatment conditions.
Period: Overall Study
Arm/Group | Arm 1: MI-CBT | Arm 2: MI-CBT+CC | Arm 3: E-TAU
Started | 60 | 60 | 60
Completed | 44 | 45 | 49
Not Completed | 16 | 15 | 11
Not completed — Lost to Follow-up | 2 | 4 | 3
Not completed — Death | 1 | 2 | 1
Not completed — Withdrawal by Subject | 10 | 8 | 4
Not completed — missing data on primary outcome | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: MI-CBT | Arm 2: MI-CBT+CC | Arm 3: E-TAU | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (12.9) | 44.9 (12.9) | 42.9 (12.8) | 42.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 55 | 55 | 55 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 55 | 55 | 57 | 167
  Unknown or Not Reported | 3 | 3 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 18 | 19 | 51
  White | 41 | 35 | 38 | 114
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 3 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Conflict Tactics Scale-Structured Interview (CTS-SI)
Description: The CTS-SI is a semi-structured interview assessing interpersonal violence (violence severity, injury and characteristics of interpersonal conflict incidents). Baseline data collection assessed the 180 days prior to enrollment, and follow-up data was collected at 3 and 6 months for the prior 90 days, and at 12 months for the past 180 days. The analysis below compares the month rate of various types of interpersonal aggression from the period pre-baseline to the monthly rate post-intervention (across all 12 months of follow-up) in the form of % difference. Means at baseline, 3 , 6 and 12 months were compared resulting in a number with no measure of dispersion. Values were calculated across all participants. There were primary aggression outcomes (overall physical aggression, injuring another person), and secondary aggression outcomes (partner physical aggression and injury, nonpartner physical aggression and injury).
Time Frame: % difference between baseline and the collapsed 3-, 6-, and 12-month follow-up data
Population: Main analyses used General Estimating Equations which accounts for missing data. Results in tables below are from bivariate analyses.
Measure: Number; unit: percentage change
Arm/Group | Arm 1: MI-CBT | Arm 2: MI-CBT+CC | Arm 3: E-TAU
Number analyzed (Participants) | 60 | 60 | 60
percentage change
  Overall physical aggression % change from baseline | -90 | -90 | -94
  Overall Injury Perpetration % change from baseline | -82 | -91 | -86
  Partner physical aggression % change from baseline | -92 | -91 | -97
  Partner injury % change from baseline | -100 | -85 | -61
  Nonpartner physical aggresion % change from baseli | -88 | -89 | -90
  Nonpartner injury % change from baseline | -76 | -93 | -99
Statistical Analysis 1: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to overall physical aggression % change from baseline; Test type: Superiority; p < 0.001, Wilcoxon Z — The threshold for significance was p < 0.05. Scores are reported stratified by whether they are less than .05 less than .01 and less than .001 respectively; Wilcoxon Z value: -4.65; Coefficient estimate = 0.82, 95% CI 2-sided [0.37 to 1.84] — E-TAU arm is the referent group
Statistical Analysis 2: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to overall injury perpetration % change from baseline; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -2.83; Coefficient Estimate = 0.62, 95% CI 2-sided [0.30 to 1.29] — E-TAU arm is the referent group
Statistical Analysis 3: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to partner physical aggression % change from baseline; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -3.31; Coefficient Estimate = 1.16, 95% CI 2-sided [0.36 to 3.77] — E-TAU arm is the referent group
Statistical Analysis 4: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to partner injury % change from baseline; Test type: Superiority; p < 0.05, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -2.26; Coefficient Estimate = 0.51, 95% CI 2-sided [0.19 to 1.38] — E-TAU arm is the referent group
Statistical Analysis 5: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to non-partner physical aggression % change from baseline; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -3.79; Coefficient Estimate = 1.22, 95% CI 2-sided [0.66 to 2.28] — E-TAU arm is the referent group
Statistical Analysis 6: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to non-partner injury % change from baseline; Test type: Superiority; p < 0.05, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -2.01; Coefficient Estimate = 0.80, 95% CI 2-sided [0.32 to 1.98] — E-TAU arm is the referent group
Statistical Analysis 7: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -4.81; Coefficient Estimate = 0.60, 95% CI 2-sided [0.25 to 1.46] — E-TAU arm is the referent group
Statistical Analysis 8: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -3.74; Coefficient Estimate = 1.05, 95% CI 2-sided [0.45 to 2.44] — E-TAU arm is the referent group
Statistical Analysis 9: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -2.59; Coefficient Estimate = 0.48, 95% CI 2-sided [0.13 to 1.78] — E-TAU arm is the referent group
Statistical Analysis 10: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p > 0.05, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -1.81; Coefficient Estimate = 0.48, 95% CI 2-sided [0.16 to 1.47] — E-TAU arm is the referent group
Statistical Analysis 11: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -4.10; Coefficient Estimate = 1.12, 95% CI 2-sided [0.60 to 2.08] — E-TAU arm is the referent group
Statistical Analysis 12: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -3.17; Coefficient Estimate = 1.09, 95% CI 2-sided [0.40 to 2.95] — E-TAU arm is the referent group
Statistical Analysis 13: Comparison: Arm 3: E-TAU; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -4.69
Statistical Analysis 14: Comparison: Arm 3: E-TAU; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to overall injury % change from baseline; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -3.32
Statistical Analysis 15: Comparison: Arm 3: E-TAU; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -2.90
Statistical Analysis 16: Comparison: Arm 3: E-TAU; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p > 0.05, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z Score: -1.02
Statistical Analysis 17: Comparison: Arm 3: E-TAU; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z Score: -4.01
Statistical Analysis 18: Comparison: Arm 3: E-TAU; Bivariate analyses examined change from baseline to follow up of primary and secondary outcomes measures using Wilcoxon sign rank tests. This test applies to overall non-partner injury % change from baseline; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 1, analysis 1]; Wilcoxon Z score: -3.21

2. Secondary Outcome: Percent Change in the Percentage of Days of Substance Use for Each Substance
Description: Data was collected via a Time-line Follow Back interview. Semi-structured interview assessing alcohol and drug use. Baseline data collection assessed the 180 days prior to enrollment, and follow-up data was collected at 3 and 6 months for the prior 90 days, and at 12 months for the past 180 days. The analysis below compares the monthly rate of various types of substance use (heavy drinking, cocaine, marijuana, and illicit) from the period pre-baseline to the monthly rate post-intervention (across all 12 months of follow-up) in the form of % difference. (% days use for each substance) Means at baseline, 3 , 6 and 12 months were compared resulting in a number with no measure of dispersion. Values were calculated across all participants.
Time Frame: % difference between baseline and the collapsed 3-, 6-, and 12-month follow-up data
Population: Main analyses used General Estimating Equations which accounts for missing data. Results in data table are from bivariate analyses.
Measure: Number; unit: percentage of change
Arm/Group | Arm 1: MI-CBT | Arm 2: MI-CBT+CC | Arm 3: E-TAU
Number analyzed (Participants) | 60 | 60 | 60
percentage of change
  Heavy Drinking % change from baseline | -68 | -59 | -55
  cocaine use % change from baseline | -83 | -86 | -56
  marijuana use % change from baseline | -40 | -42 | -44
  Overall illicit drug use % change from baseline | -52 | -50 | -57
Statistical Analysis 1: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of substance use outcomes measures using Wilcoxon sign rank tests. This test applies to heavy drinking % change from baseline; Test type: Superiority; p < 0.001, Wilcoxon Z — The threshold for significance was p<0.05. Scores are reported stratified by whether they are less than 0.05, less than 0.01, and less than 0.001; Wilcoxon Z value: -3.52; Coefficient estimate = 0.95, 95% CI 2-sided [0.62 to 1.47] — E-TAU arm is the referent group
Statistical Analysis 2: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of substance use outcomes measures using Wilcoxon sign rank tests. This test applies to cocaine use % change from baseline; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -2.98; coefficient estimate = 0.49, 95% CI 2-sided [0.18 to 1.32] — E-TAU arm is the referent group
Statistical Analysis 3: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of substance use outcomes measures using Wilcoxon sign rank tests. This test applies to marijuana use % change from baseline; Test type: Superiority; p < 0.05, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -2.13; coefficient estimate = 0.85, 95% CI 2-sided [0.4 to 1.8] — E-TAU arm is the referent group
Statistical Analysis 4: Comparison: Arm 1: MI-CBT; Bivariate analyses examined change from baseline to follow up of substance use outcomes measures using Wilcoxon sign rank tests. This test applies to illicit drug use % change from baseline; Test type: Superiority; p < 0.05, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -2.48; coefficient estimate = 0.84, 95% CI 2-sided [0.54 to 1.32] — E-TAU arm is the referent group
Statistical Analysis 5: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -4.94; coefficient estimate = 1.15, 95% CI 2-sided [0.78 to 1.71] — E-TAU arm is the referent group
Statistical Analysis 6: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.05, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -2.56; coefficient estimate = 0.61, 95% CI 2-sided [0.17 to 2.16] — E-TAU arm is the referent group
Statistical Analysis 7: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.01, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -2.86; coefficient estimate = 1.18, 95% CI 2-sided [0.57 to 2.44] — E-TAU arm is the referent group
Statistical Analysis 8: Comparison: Arm 2: MI-CBT+CC; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -3.51; coefficient estimate = 0.95, 95% CI 2-sided [0.61 to 1.48] — E-TAU arm is the referent group
Statistical Analysis 9: Comparison: Arm 3: E-TAU; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -4.65
Statistical Analysis 10: Comparison: Arm 3: E-TAU; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p > 0.05, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -1.45
Statistical Analysis 11: Comparison: Arm 3: E-TAU; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p > 0.05, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -1.5
Statistical Analysis 12: Comparison: Arm 3: E-TAU; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p < 0.05, Wilcoxon Z — [p-value comment as in outcome 2, analysis 1]; Wilcoxon Z value: -2.58

ADVERSE EVENTS:
Description: In the event of participant death, cause of death is unknown.
Arm/Group | Arm 1: MI-CBT | Arm 2: MI-CBT+CC | Arm 3: E-TAU
All-Cause Mortality (participants affected / at risk) | 1/60 | 2/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/60 | 1/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: MI-CBT (N=60) | Arm 2: MI-CBT+CC (N=60) | Arm 3: E-TAU (N=60)
Participant Death (Social circumstances) | 1 (1) | 2 (2) | 1 (1) — There were 4 serious adverse events involving participant deaths. These were immediately reported to our IRB, and none of the events was considered to be study related.

LIMITATIONS AND CAVEATS:
We fell short of recruitment goal of 210 participants and had a low number of women per group. Rates of aggression at each follow-up were very low so we collapsed across the 3,6 & 12 month follow-ups when examining changes from baseline to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes